CLINICAL TRIAL: NCT04159805
Title: A Phase 2, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Efficacy of TAK-079 in Patients With Generalized Myasthenia Gravis
Brief Title: A Study of TAK-079 in People With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-079-1005; 2019-003383-47 (EudraCT Number)
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Myasthenia Gravis
Keywords: Drug therapy
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-079 Placebo-matching (Placebo Comparator): TAK-079 placebo-matching injection, subcutaneously (SC), once weekly in combination with standard background therapy for 8 weeks.
  Interventions: Drug: TAK-079 Placebo
- TAK-079 300 mg (Experimental): TAK-079 300 mg injection, SC, once weekly in combination with standard background therapy for 8 weeks.
  Interventions: Drug: TAK-079
- TAK-079 600 mg (Experimental): TAK-079 600 mg injection, SC, once weekly in combination with standard background therapy for 8 weeks.
  Interventions: Drug: TAK-079

INTERVENTIONS:
Drug: TAK-079 — TAK-079 subcutaneous injection
  Other Names: Mezagitamab
  Arms: TAK-079 300 mg; TAK-079 600 mg
Drug: TAK-079 Placebo — TAK-079 placebo-matching subcutaneous injection
  Arms: TAK-079 Placebo-matching

SUMMARY:
Myasthenia gravis is an autoimmune condition that causes muscle weakness. Autoimmune means the body makes antibodies that attack its own cells and tissues. These types of antibodies are also known as autoantibodies. People with generalized myasthenia gravis have a weakness in many muscles.

TAK-079 is a medicine to help people with generalized myasthenia gravis.

The main aim of this study is to check if people with generalized myasthenia gravis have side effects from 2 doses of TAK-079. Other aims are to learn if TAK-079 improves their clinical condition and lowers their autoantibody levels.

At the first visit, the study doctor will check if each person can take part. For those who can take part, participants will continue with their standard medicines for this condition during the study. Each participant will have a check-up by the study doctor.

Then, the participants will have 1 of 3 treatments:

* A low dose of TAK-079.
* A high dose of TAK-079.
* A placebo. In this study, a placebo looks like TAK-079 but does not have any medicine in it.

Participants will not know which treatment they received, nor will their study doctors. This is to help make sure the results are more reliable.

For each treatment, participants will receive injections just under the skin, once a week for 8 weeks. The study doctors will check for side effects from the study treatments. The study doctors can stop or delay the injections in each participant if needed.

Then, the study doctors will continue to check for side effects for up to 24 weeks after treatment. They will also check the clinical condition of the participants, including their autoantibody levels.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune disorder in which autoantibodies, such as those targeting the nicotinic acetylcholine receptor (AChR) or muscle specific kinase (MuSK), interfere with neuromuscular transmission, resulting in fatigue and weakness.

The drug being tested in this study is called TAK-079. TAK-079 is being tested to treat people who have generalized myasthenia gravis.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of Myasthenia Gravis (MG) supported by a positive serologic test for anti-AChR or anti-MuSK antibodies at screening.
2. Myasthenia Gravis Foundation of America (MGFA) clinical classification II to IV at screening.
3. Myasthenia Gravis Activities of Daily Living (MG-ADL) total score of 6 or greater at screening, with at least 4 points attributed to nonocular items.
4. If receiving immunosuppressive drugs (ie, mycophenolate mofetil, methotrexate, cyclosporine, tacrolimus, cyclophosphamide), therapy must be ongoing for at least 6 months, with stable dosing ongoing for at least 3 months before screening. Participants receiving azathioprine must be on a stable dose for at least 6 months before screening.
5. If receiving oral corticosteroids, therapy must be ongoing for at least 3 months, with a stable dose at least 1 month before screening. Corticosteroids, including dexamethasone, must be given as oral, daily or every-other-day therapy, as opposed to pulse therapy.
6. If receiving cholinesterase inhibitors, therapy with a stable dose is required at least 2 weeks before screening.
7. The doses of concomitant standard background therapy must be expected to remain stable throughout the study unless dose reduction is required due to toxicities. Allowed background therapy is defined as no more than a cholinesterase inhibitor ± corticosteroid ± 1 steroid-sparing immunosuppressive drug (limited to azathioprine, mycophenolate mofetil, methotrexate, cyclosporine, tacrolimus, or cyclophosphamide). Participants must be on at least one allowed background medication.

Main Exclusion Criteria:

1. Presence of a thymoma (previous history of a fully encapsulated thymoma removed ≥ 12 months before screening is allowed) or history of invasive thymic malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥ 5 years before screening.
2. History of thymectomy within 12 months before screening.
3. MGFA class I or V.
4. Received intravenous immunoglobulin (IVIg), subcutaneous immunoglobulin (SCIg), or plasmapheresis/plasma exchange within 4 weeks before screening, or an expectation that any therapy besides the participants standard background therapies may be used for treatment of MG (eg, a rescue therapy) between screening and dosing.
5. Chronic obstructive pulmonary disease (COPD) or asthma with a pre-bronchodilatory forced expiratory volume in 1 second (FEV1) <50% of predicted normal.

   Note: FEV1 testing is required for participants suspected of having COPD or asthma.
6. Received rituximab, belimumab, eculizumab, or any monoclonal antibody for immunomodulation within 6 months before first dosing. Participants with prior exposure to rituximab must have CD19 counts within the normal range at screening.
7. Known autoimmune disease other than MG that could interfere with the course and conduct of the study.
8. Received a live vaccine within 4 weeks before screening or has any live vaccination planned during the study.
9. Opportunistic infection ≤12 weeks before initial study dosing or currently receiving treatment for a chronic opportunistic infection, such as tuberculosis (TB), pneumocystis pneumonia, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria. A mild, localized herpes simplex infection within 12 weeks of study dosing is allowed, as long as the lesion has resolved without systemic therapy prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (49):
- United States (26):
  - The University of Arizona Medical Center, Tucson, Arizona
  - Stanford Neuroscience Health Center, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Neurology Associates PA, Maitland, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - Augusta University, Augusta, Georgia
  - Consultants In Neurology, Northbrook, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Neurology and Sleep Disorders Clinic, Columbia, Missouri
  - Hospital For Special Surgery, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas HealthCare System Neurosciences Institute-Neurology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Austin Neuromuscular Center, Austin, Texas
  - The University of Texas South Western Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants PA, Round Rock, Texas
  - Center for Neurological Disorders, Milwaukee, Wisconsin
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Canada (3):
  - The Governors of the University of Calgary, Calgary, Alberta
  - Vancouver General Hospital (VGH), Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
- Italy (5):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS AOU San Martino, Genova
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Sant'andrea, Rome
- Poland (4):
  - Neurocentrum Bydgoszcz sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Neurologii Klinicznej Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne NeuroProtect, Warsaw
  - Centrum Medyczne Warszawa - PRATIA - PPDS, Warsaw
- Serbia (3):
  - Clinical Center of Serbia - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Nis, Niš
- Spain (8):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in the United States, Spain, Poland, Serbia, and Canada from 14 January 2020 to 12 July 2022.
Pre-assignment Details: Participants with a diagnosis of Myasthenia Gravis (MG) were enrolled in 1:1:1 ratio to receive TAK-079 matching placebo, TAK-079 300 mg or TAK-079 600 mg in combination with standard background therapy.
Period: Overall Study
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Started | 12 | 12 | 12
Completed | 12 | 10 | 10
Not Completed | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Groups:
- TAK-079 Placebo-matching: TAK-079 placebo-matching injection, SC, once weekly in combination with standard background therapy for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (18.03) | 45.3 (12.47) | 56.3 (14.42) | 49.4 (15.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 7 | 22
  Male | 3 | 6 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 9 | 12 | 11 | 32
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 10 | 12 | 11 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 1 | 2
  Poland | 1 | 2 | 2 | 5
  Serbia | 5 | 7 | 5 | 17
  Spain | 3 | 0 | 1 | 4
  United States | 3 | 2 | 3 | 8
Height [Mean (Standard Deviation); unit: cm] | 164.67 (9.435) | 175.39 (8.911) | 171.38 (10.910) | 170.48 (10.511)
Weight [Mean (Standard Deviation); unit: kg] | 85.11 (25.607) | 86.28 (21.132) | 88.38 (25.672) | 86.59 (23.568)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=[weight(kg) / height(m)^2].
  kg/m^2 | 31.33 (8.867) | 27.74 (4.852) | 30.22 (9.315) | 29.76 (7.855)
Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Participant-reported scale to assess MG symptoms to evaluate capacity to perform activities of daily living. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 24; the higher score indicates greater functional impairment and disability.
  score on a scale | 7.9 (1.78) | 9.3 (2.49) | 8.4 (2.23) | 8.5 (2.20)
Quantitative Myasthenia Gravis (QMG) Scale Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Physician-reported scale to assess MG disease severity by quantifying several body functions by physical exam. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 39; the higher score indicates greater disease burden.
  score on a scale | 11.4 (5.21) | 12.9 (6.47) | 12.8 (4.26) | 12.4 (5.28)
Myasthenia Gravis Composite (MGC) Scale Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — An assessment scale of MG disease activity based on a combination of participant- and physician-reported items. Items are scored based on 4 potential levels of impact: normal, mild, moderate, or severe with a total score of 0 to 50; the higher score indicates worse MG disease activity.
  score on a scale | 14.7 (5.80) | 16.8 (6.58) | 15.3 (6.00) | 15.6 (6.03)
Revised 15-item Myasthenia Gravis Quality of Life Scale (MG-QoL15r) Scale Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — A participant-reported score that assesses the participant's perception of impairment and disability and the degree to which the patient tolerates disease manifestations. Each question is graded on a 3-point scale from 0=normal to 2=severe with a total score of 0 to 30; the higher score indicates worse MG disease activity.
  score on a scale | 11.5 (4.15) | 17.1 (6.76) | 13.9 (4.72) | 14.2 (5.67)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Grade 3 or Higher TEAEs, and Adverse Event (AE) Leading to TAK-079 Discontinuation
Description: AE is defined as any untoward medical occurrence in clinical investigation participant administered drug; it does not necessarily have to have causal relationship with this treatment. TEAE is defined as AE with onset that occurs after receiving study drug. SAE is an adverse event resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Severity of TEAEs was graded using National cancer institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 definitions of Grade 1 through Grade 5 wherein Grade 1=mild symptoms, Grade 2=moderate symptoms, Grade 3=Severe or medically significant but not immediately life-threatening, Grade 4=life-threatening consequences and Grade 5=death related to AEs. Percentages are rounded off to whole number at single decimal.
Time Frame: From signing the informed consent form up to end of long-term follow-up (up to Week 32)
Population: Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants
  TEAE | 66.7 | 75.0 | 91.7
  SAE | 8.3 | 8.3 | 8.3
  Grade 3 or Higher TEAEs | 16.7 | 8.3 | 8.3
  AE Leading to TAK-079 Discontinuation | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Change From Baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale Score
Description: Participant-reported scale to assess MG symptoms to evaluate capacity to perform activities of daily living. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 24; the higher score indicates greater functional impairment and disability. Negative change indicates improvement. Mixed-effects model for repeated measures (MMRM) was used for the analysis.
Time Frame: Baseline up to Week 32
Population: Full Analysis Set included all randomized participants who had baseline and at least 1 post-baseline efficacy assessment. Number analyzed is the number of participants available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Change From Baseline at Week 4 | -2.8 (2.67) | -2.5 (2.47) | -1.8 (1.66)
  Change From Baseline at Week 6: number analyzed (Participants) | 12 | 11 | 11
  Change From Baseline at Week 6 | -4.0 (2.73) | -4.2 (2.64) | -2.3 (2.15)
  Change From Baseline at Week 8: number analyzed (Participants) | 12 | 11 | 12
  Change From Baseline at Week 8 | -3.8 (2.80) | -4.3 (3.10) | -2.0 (3.16)
  Change From Baseline at Week 10: number analyzed (Participants) | 11 | 11 | 11
  Change From Baseline at Week 10 | -4.0 (3.52) | -5.0 (2.41) | -2.0 (2.79)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 11 | 12
  Change From Baseline at Week 12 | -4.2 (3.19) | -4.2 (2.56) | -2.5 (2.68)
  Change From Baseline at Week 14: number analyzed (Participants) | 11 | 10 | 10
  Change From Baseline at Week 14 | -4.0 (4.38) | -4.8 (2.20) | -2.0 (3.30)
  Change From Baseline at Week 16: number analyzed (Participants) | 10 | 10 | 10
  Change From Baseline at Week 16 | -4.1 (3.21) | -4.3 (2.79) | -3.1 (3.48)
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 8 | 11
  Change From Baseline at Week 20 |  | -3.9 (3.60) | -2.9 (3.11)
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 9 | 9
  Change From Baseline at Week 24 |  | -4.1 (3.62) | -3.0 (3.57)
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 10 | 9
  Change From Baseline at Week 28 |  | -3.9 (3.96) | -3.1 (3.37)
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 9 | 8
  Change From Baseline at Week 32 |  | -2.3 (4.61) | -2.8 (3.99)
Statistical Analysis 1: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.772, MMRM — From MMRM analysis over all post-baseline visits, with the change from baseline as the outcome, treatment group, visit, and treatment-by-visit interaction as factors, and adjusted by baseline value and baseline-by-visit interaction; Difference in Least Square (LS) Mean = 0.29, 95% CI 2-sided [-1.72 to 2.30]
Statistical Analysis 2: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.299, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.01, 95% CI 2-sided [-0.94 to 2.97]
Statistical Analysis 3: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.924, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.11, 95% CI 2-sided [-2.34 to 2.13]
Statistical Analysis 4: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.091, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.86, 95% CI 2-sided [-0.32 to 4.04]
Statistical Analysis 5: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.887, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.18, 95% CI 2-sided [-2.82 to 2.45]
Statistical Analysis 6: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.162, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.80, 95% CI 2-sided [-0.76 to 4.36]
Statistical Analysis 7: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.784, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.36, 95% CI 2-sided [-3.01 to 2.29]
Statistical Analysis 8: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.166, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.79, 95% CI 2-sided [-0.79 to 4.37]
Statistical Analysis 9: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.724, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.42, 95% CI 2-sided [-1.98 to 2.82]
Statistical Analysis 10: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.124, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.81, 95% CI 2-sided [-0.52 to 4.14]
Statistical Analysis 11: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.856, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.29, 95% CI 2-sided [-2.91 to 3.48]
Statistical Analysis 12: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.292, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.64, 95% CI 2-sided [-1.48 to 4.76]
Statistical Analysis 13: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.944, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.11, 95% CI 2-sided [-3.14 to 3.37]
Statistical Analysis 14: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.589, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.85, 95% CI 2-sided [-2.33 to 4.02]

3. Secondary Outcome: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Scale Score
Description: Physician-reported scale to assess MG disease severity by quantifying several body functions by physical exam. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 39; the higher score indicates greater disease burden. Negative change indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline up to Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Change From Baseline at Week 4 | -1.0 (2.34) | -2.0 (2.70) | -0.2 (2.89)
  Change From Baseline at Week 6: number analyzed (Participants) | 11 | 12 | 12
  Change From Baseline at Week 6 | -0.9 (1.76) | -2.5 (3.24) | -1.3 (3.10)
  Change From Baseline at Week 8: number analyzed (Participants) | 12 | 11 | 11
  Change From Baseline at Week 8 | -1.0 (2.30) | -3.4 (3.35) | -0.9 (3.27)
  Change From Baseline at Week 10: number analyzed (Participants) | 11 | 11 | 11
  Change From Baseline at Week 10 | -1.4 (2.87) | -3.2 (3.09) | -0.7 (4.03)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 11 | 12
  Change From Baseline at Week 12 | -2.8 (2.68) | -3.9 (2.55) | -0.8 (3.51)
  Change From Baseline at Week 14: number analyzed (Participants) | 11 | 10 | 10
  Change From Baseline at Week 14 | -1.9 (3.11) | -3.5 (2.51) | 0.6 (4.65)
  Change From Baseline at Week 16: number analyzed (Participants) | 10 | 10 | 10
  Change From Baseline at Week 16 | -1.2 (3.22) | -3.3 (3.43) | -0.3 (4.81)
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 8 | 11
  Change From Baseline at Week 20 |  | -1.9 (3.56) | -0.5 (4.27)
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 9 | 9
  Change From Baseline at Week 24 |  | -2.2 (4.47) | -0.6 (3.78)
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 10 | 9
  Change From Baseline at Week 28 |  | -1.7 (3.80) | -0.8 (4.52)
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 9 | 8
  Change From Baseline at Week 32 |  | -0.7 (4.27) | -0.1 (4.79)
Statistical Analysis 1: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.406, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.93, 95% CI 2-sided [-3.17 to 1.31]
Statistical Analysis 2: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.418, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.90, 95% CI 2-sided [-1.34 to 3.14]
Statistical Analysis 3: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.463, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.94, 95% CI 2-sided [-3.53 to 1.65]
Statistical Analysis 4: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.936, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.10, 95% CI 2-sided [-2.70 to 2.49]
Statistical Analysis 5: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.170, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -1.80, 95% CI 2-sided [-4.41 to 0.82]
Statistical Analysis 6: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.687, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.52, 95% CI 2-sided [-2.10 to 3.13]
Statistical Analysis 7: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.374, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -1.24, 95% CI 2-sided [-4.05 to 1.57]
Statistical Analysis 8: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.478, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.99, 95% CI 2-sided [-1.82 to 3.80]
Statistical Analysis 9: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.690, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.51, 95% CI 2-sided [-3.12 to 2.09]
Statistical Analysis 10: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.106, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 2.12, 95% CI 2-sided [-0.48 to 4.71]
Statistical Analysis 11: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.547, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.89, 95% CI 2-sided [-3.89 to 2.12]
Statistical Analysis 12: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.144, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 2.19, 95% CI 2-sided [-0.81 to 5.18]
Statistical Analysis 13: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.431, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -1.37, 95% CI 2-sided [-4.91 to 2.17]
Statistical Analysis 14: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.488, MMRM; Difference in LS Mean = 1.20, 95% CI 2-sided [-2.34 to 4.74]

4. Secondary Outcome: Change From Baseline in Myasthenia Gravis Composite (MGC) Scale Score
Description: An assessment scale of MG disease activity based on a combination of participant- and physician-reported items. Items are scored based on 4 potential levels of impact: normal, mild, moderate, or severe with a total score of 0 to 50; the higher score indicates worse MG disease activity. Negative change indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline up to Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Change From Baseline at Week 4 | -4.2 (3.69) | -4.9 (3.82) | -1.1 (5.92)
  Change From Baseline at Week 6: number analyzed (Participants) | 12 | 11 | 11
  Change From Baseline at Week 6 | -7.3 (4.29) | -6.1 (5.24) | -4.9 (4.74)
  Change From Baseline at Week 8: number analyzed (Participants) | 11 | 11 | 12
  Change From Baseline at Week 8 | -5.5 (4.03) | -7.4 (4.63) | -2.4 (6.10)
  Change From Baseline at Week 10: number analyzed (Participants) | 11 | 11 | 11
  Change From Baseline at Week 10 | -7.8 (5.86) | -7.6 (5.07) | -2.6 (6.55)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 11 | 12
  Change From Baseline at Week 12 | -7.3 (5.00) | -8.5 (3.11) | -5.1 (5.11)
  Change From Baseline at Week 14: number analyzed (Participants) | 11 | 10 | 10
  Change From Baseline at Week 14 | -6.1 (6.52) | -9.7 (3.83) | -0.9 (8.25)
  Change From Baseline at Week 16: number analyzed (Participants) | 10 | 10 | 10
  Change From Baseline at Week 16 | -6.6 (4.95) | -9.2 (5.18) | -2.9 (6.45)
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 8 | 11
  Change From Baseline at Week 20 |  | -7.3 (5.20) | -2.6 (7.21)
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 9 | 9
  Change From Baseline at Week 24 |  | -7.1 (5.78) | -3.3 (7.30)
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 10 | 9
  Change From Baseline at Week 28 |  | -5.6 (6.40) | -4.1 (7.59)
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 9 | 8
  Change From Baseline at Week 32 |  | -3.4 (8.13) | -2.5 (8.07)
Statistical Analysis 1: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.855, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.34, 95% CI 2-sided [-4.14 to 3.45]
Statistical Analysis 2: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.093, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 3.19, 95% CI 2-sided [-0.56 to 6.95]
Statistical Analysis 3: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.410, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.80, 95% CI 2-sided [-2.61 to 6.20]
Statistical Analysis 4: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.154, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 3.13, 95% CI 2-sided [-1.25 to 7.50]
Statistical Analysis 5: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.662, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.94, 95% CI 2-sided [-5.29 to 3.41]
Statistical Analysis 6: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.130, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 3.26, 95% CI 2-sided [-1.02 to 7.54]
Statistical Analysis 7: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.586, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.27, 95% CI 2-sided [-3.44 to 5.98]
Statistical Analysis 8: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.039, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 4.93, 95% CI 2-sided [0.26 to 9.60]
Statistical Analysis 9: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.909, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.22, 95% CI 2-sided [-4.03 to 3.60]
Statistical Analysis 10: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.158, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 2.65, 95% CI 2-sided [-1.09 to 6.40]
Statistical Analysis 11: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.764, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -0.88, 95% CI 2-sided [-6.80 to 5.05]
Statistical Analysis 12: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.080, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 5.20, 95% CI 2-sided [-0.67 to 11.06]
Statistical Analysis 13: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.677, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -1.01, 95% CI 2-sided [-5.98 to 3.95]
Statistical Analysis 14: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.055, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 4.81, 95% CI 2-sided [-0.10 to 9.73]

5. Secondary Outcome: Change From Baseline in Revised 15-item Myasthenia Gravis Quality of Life Scale (MG-QoL15r) Scale Score
Description: A participant-reported score that assesses the participant's perception of impairment and disability and the degree to which the participant tolerates disease manifestations. Each question is graded on a 3-point scale from 0=normal to 2=severe with a total score of 0 to 30; the higher score indicates worse MG disease activity. Negative change indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline up to Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Change From Baseline at Week 4 | -3.1 (3.85) | -3.9 (4.46) | -3.2 (4.43)
  Change From Baseline at Week 6: number analyzed (Participants) | 12 | 11 | 11
  Change From Baseline at Week 6 | -4.3 (4.11) | -5.8 (6.00) | -3.4 (3.53)
  Change From Baseline at Week 8: number analyzed (Participants) | 12 | 11 | 12
  Change From Baseline at Week 8 | -3.2 (4.00) | -5.6 (6.53) | -3.3 (3.74)
  Change From Baseline at Week 10: number analyzed (Participants) | 11 | 11 | 11
  Change From Baseline at Week 10 | -2.5 (6.12) | -6.3 (6.07) | -3.9 (3.70)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 11 | 12
  Change From Baseline at Week 12 | -2.5 (5.32) | -6.1 (7.25) | -4.1 (4.40)
  Change From Baseline at Week 14: number analyzed (Participants) | 11 | 10 | 10
  Change From Baseline at Week 14 | -2.0 (7.06) | -6.4 (6.98) | -0.9 (5.49)
  Change From Baseline at Week 16: number analyzed (Participants) | 10 | 10 | 10
  Change From Baseline at Week 16 | -3.8 (4.44) | -5.8 (6.83) | -2.3 (6.43)
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 8 | 11
  Change From Baseline at Week 20 |  | -3.3 (7.01) | -4.7 (5.48)
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 8 | 9
  Change From Baseline at Week 24 |  | -7.1 (7.95) | -3.8 (5.31)
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 10 | 8
  Change From Baseline at Week 28 |  | -4.8 (10.36) | -4.0 (6.16)
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 9 | 8
  Change From Baseline at Week 32 |  | -6.2 (7.31) | -2.4 (4.78)
Statistical Analysis 1: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.780, MMRM — From a MMRM analysis over all post-baseline visits, with the change from baseline as the outcome, treatment group, visit, and treatment-by-visit interaction as factors, and adjusted by baseline value and baseline-by-visit interaction; Difference in LS Mean = 0.52, 95% CI 2-sided [-3.23 to 4.27]
Statistical Analysis 2: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.771, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 0.50, 95% CI 2-sided [-2.99 to 3.99]
Statistical Analysis 3: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.984, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -0.04, 95% CI 2-sided [-4.22 to 4.14]
Statistical Analysis 4: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.213, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 2.44, 95% CI 2-sided [-1.47 to 6.35]
Statistical Analysis 5: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.371, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -1.97, 95% CI 2-sided [-6.40 to 2.45]
Statistical Analysis 6: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.956, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 0.11, 95% CI 2-sided [-4.01 to 4.23]
Statistical Analysis 7: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.641, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -1.06, 95% CI 2-sided [-5.65 to 3.53]
Statistical Analysis 8: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.876, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -0.33, 95% CI 2-sided [-4.61 to 3.95]
Statistical Analysis 9: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.458, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -1.86, 95% CI 2-sided [-6.91 to 3.18]
Statistical Analysis 10: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.769, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -0.68, 95% CI 2-sided [-5.37 to 4.00]
Statistical Analysis 11: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.699, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = -1.14, 95% CI 2-sided [-7.07 to 4.80]
Statistical Analysis 12: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 14; Test type: Superiority; p = 0.687, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 1.10, 95% CI 2-sided [-4.41 to 6.62]
Statistical Analysis 13: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.944, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 0.20, 95% CI 2-sided [-5.55 to 5.95]
Statistical Analysis 14: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 16; Test type: Superiority; p = 0.351, MMRM — [p-value comment as in outcome 5, analysis 1]; Difference in LS Mean = 2.48, 95% CI 2-sided [-2.87 to 7.83]

6. Secondary Outcome: Change From Baseline in Anti-acetylcholine Receptor (AChR) Antibody Levels
Description: Clinical laboratory evaluations of anti-AChR antibodies were tested to monitor disease activity. MMRM was used for the analysis.
Time Frame: Baseline up to Week 32
Population: Full Analysis Set included all randomized participants who had baseline and at least 1 post-baseline efficacy assessment. Overall number analyzed is the number of participants available for analyses. Number analyzed is the number of participants available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 11 | 10 | 12
nmol/L
  Change From Baseline at Week 2 | 6.300 (25.3514) | -19.452 (50.5551) | -3.450 (5.7767)
  Change From Baseline at Week 3 | -3.989 (22.9732) | -14.821 (44.4776) | 2.509 (17.5221)
  Change From Baseline at Week 4 | 0.976 (11.7759) | -24.253 (51.2627) | 13.680 (87.1669)
  Change From Baseline at Week 5 | -8.199 (13.9571) | -32.251 (58.3701) | -9.831 (26.2188)
  Change From Baseline at Week 6: number analyzed (Participants) | 11 | 9 | 11
  Change From Baseline at Week 6 | -19.152 (49.2221) | -27.518 (52.6672) | -2.148 (23.2543)
  Change From Baseline at Week 7: number analyzed (Participants) | 11 | 9 | 11
  Change From Baseline at Week 7 | -11.235 (26.2159) | -33.261 (56.3495) | -9.882 (16.2972)
  Change From Baseline at Week 8: number analyzed (Participants) | 10 | 9 | 12
  Change From Baseline at Week 8 | 7.731 (27.8994) | -39.386 (72.3110) | -5.668 (10.4493)
  Change From Baseline at Week 10: number analyzed (Participants) | 10 | 9 | 11
  Change From Baseline at Week 10 | -37.473 (120.9186) | -37.083 (60.8092) | -6.654 (7.8236)
  Change From Baseline at Week 12: number analyzed (Participants) | 10 | 9 | 12
  Change From Baseline at Week 12 | -0.832 (31.0318) | -38.430 (64.4594) | -7.827 (11.2120)
  Change From Baseline at Week 14: number analyzed (Participants) | 9 | 8 | 10
  Change From Baseline at Week 14 | 12.729 (49.8823) | -40.771 (74.3624) | -8.058 (15.8407)
  Change From Baseline at Week 16: number analyzed (Participants) | 7 | 8 | 10
  Change From Baseline at Week 16 | 3.501 (9.8729) | -49.843 (77.6316) | -4.909 (8.8478)
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 7 | 11
  Change From Baseline at Week 20 |  | -52.217 (83.1537) | -4.378 (7.7297)
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 7 | 9
  Change From Baseline at Week 24 |  | -43.079 (77.4438) | -4.802 (10.5639)
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 8 | 9
  Change From Baseline at Week 28 |  | -73.786 (111.0044) | -6.044 (11.3755)
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 7 | 8
  Change From Baseline at Week 32 |  | -51.296 (67.3437) | -5.485 (11.8380)
Statistical Analysis 1: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 2; Test type: Superiority; p = 0.090, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -27.90, 95% CI 2-sided [-60.18 to 4.38]
Statistical Analysis 2: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 2; Test type: Superiority; p = 0.328, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -15.77, 95% CI 2-sided [-47.50 to 15.96]
Statistical Analysis 3: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 3; Test type: Superiority; p = 0.441, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -12.65, 95% CI 2-sided [-44.94 to 19.63]
Statistical Analysis 4: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 3; Test type: Superiority; p = 0.931, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 1.39, 95% CI 2-sided [-30.33 to 33.12]
Statistical Analysis 5: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.087, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -28.18, 95% CI 2-sided [-60.46 to 4.11]
Statistical Analysis 6: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 4; Test type: Superiority; p = 0.783, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 4.44, 95% CI 2-sided [-27.29 to 36.16]
Statistical Analysis 7: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 5; Test type: Superiority; p = 0.077, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -29.08, 95% CI 2-sided [-61.36 to 3.21]
Statistical Analysis 8: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 5; Test type: Superiority; p = 0.330, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -15.72, 95% CI 2-sided [-47.45 to 16.00]
Statistical Analysis 9: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 6; Test type: Superiority; p = 0.400, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -14.14, 95% CI 2-sided [-47.19 to 18.91]
Statistical Analysis 10: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 6; Test type: Superiority; p = 1.000, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = 0.00, 95% CI 2-sided [-32.18 to 32.19]
Statistical Analysis 11: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 7; Test type: Superiority; p = 0.117, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -26.47, 95% CI 2-sided [-59.64 to 6.69]
Statistical Analysis 12: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 7; Test type: Superiority; p = 0.436, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -12.75, 95% CI 2-sided [-44.94 to 19.44]
Statistical Analysis 13: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 8; Test type: Superiority — From MMRM analysis over all post-baseline visits, with the change from baseline as the outcome, treatment group, visit, and treatment-by-visit interaction as factors, and adjusted by baseline value and baseline-by-visit interaction; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -47.91, 95% CI 2-sided [-81.54 to -14.29]
Statistical Analysis 14: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 8; Test type: Superiority; p = 0.215, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -20.48, 95% CI 2-sided [-52.92 to 11.95]
Statistical Analysis 15: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.815, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -3.97, 95% CI 2-sided [-37.34 to 29.40]
Statistical Analysis 16: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Change From Baseline at Week 10; Test type: Superiority; p = 0.794, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -4.31, 95% CI 2-sided [-36.84 to 28.22]
Statistical Analysis 17: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.033, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -36.78, 95% CI 2-sided [-70.48 to -3.08]
Statistical Analysis 18: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Week 12; Test type: Superiority; p = 0.513, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -10.79, 95% CI 2-sided [-43.26 to 21.67]
Statistical Analysis 19: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Week 14; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -56.21, 95% CI 2-sided [-91.69 to -20.73]
Statistical Analysis 20: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Week 14; Test type: Superiority; p = 0.036, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -36.94, 95% CI 2-sided [-71.39 to -2.48]
Statistical Analysis 21: Comparison: TAK-079 Placebo-matching vs TAK-079 300 mg; Week 16; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -62.98, 95% CI 2-sided [-100.64 to -25.31]
Statistical Analysis 22: Comparison: TAK-079 Placebo-matching vs TAK-079 600 mg; Week 16; Test type: Superiority; p = 0.130, MMRM — [p-value comment as in outcome 2, analysis 1]; Difference in LS Mean = -28.81, 95% CI 2-sided [-66.12 to 8.51]

7. Secondary Outcome: Change From Baseline in Anti- Muscle-specific Tyrosine Kinase (MuSK) Titer Levels
Description: Clinical laboratory evaluations of anti-MuSK antibodies were tested to monitor disease activity. Data is reported for participants who were positive for anti-MuSK antibodies at baseline.
Time Frame: Baseline up to Week 32
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 1 | 2 | 0
titer
  Change From Baseline at Week 2 | 0.0 (NA) — Standard deviation (SD) was not estimable for 1 participant. | -160.0 (226.27) |
  Change From Baseline at Week 3 | 0.0 (NA) — SD was not estimable for 1 participant. | -200.0 (169.71) |
  Change From Baseline at Week 4 | 0.0 (NA) — SD was not estimable for 1 participant. | -240.0 (339.41) |
  Change From Baseline at Week 5 | 0.0 (NA) — SD was not estimable for 1 participant. | -240.0 (339.41) |
  Change From Baseline at Week 6 | 0.0 (NA) — SD was not estimable for 1 participant. | -240.0 (339.41) |
  Change From Baseline at Week 7 | 0.0 (NA) — SD was not estimable for 1 participant. | -240.0 (339.41) |
  Change From Baseline at Week 8 | 0.0 (NA) — SD was not estimable for 1 participant. | -280.0 (395.98) |
  Change From Baseline at Week 10 | 0.0 (NA) — SD was not estimable for 1 participant. | -280.0 (395.98) |
  Change From Baseline at Week 12 | 0.0 (NA) — SD was not estimable for 1 participant. | -300.0 (424.26) |
  Change From Baseline at Week 14 | 0.0 (NA) — SD was not estimable for 1 participant. | -300.0 (424.26) |
  Change From Baseline at Week 16 | 0.0 (NA) — SD was not estimable for 1 participant. | -300.0 (424.26) |
  Change From Baseline at Week 20: number analyzed (Participants) | 0 | 1 | 0
  Change From Baseline at Week 20 |  | 0.0 (NA) — SD was not estimable for 1 participant. |
  Change From Baseline at Week 24: number analyzed (Participants) | 0 | 2 | 0
  Change From Baseline at Week 24 |  | -310.0 (438.41) |
  Change From Baseline at Week 28: number analyzed (Participants) | 0 | 2 | 0
  Change From Baseline at Week 28 |  | -310.0 (438.41) |
  Change From Baseline at Week 32: number analyzed (Participants) | 0 | 2 | 0
  Change From Baseline at Week 32 |  | -310.0 (438.41) |

8. Secondary Outcome: Percentage of Participants With 2-point Reduction in MG-ADL Total Score
Description: The percentage of responders with at least a 2-point reduction in MG-ADL total score from baseline is reported. MG-ADL is a participant-reported scale to assess MG symptoms to evaluate capacity to perform activities of daily living. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 24; the higher score indicates greater functional impairment and disability. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: At Weeks 4, 6, 8, 10, 12, 14, 16, 20, 24, 28 and 32
Population: Full Analysis Set included all randomized participants who had baseline and at least 1 post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants
  Week 4 | 50.00 | 75.00 | 58.33
  Week 6 | 91.67 | 75.00 | 58.33
  Week 8 | 83.33 | 66.67 | 66.67
  Week 10 | 83.33 | 83.33 | 50.00
  Week 12 | 75.00 | 75.00 | 50.00
  Week 14 | 66.67 | 75.00 | 50.00
  Week 16 | 66.67 | 66.67 | 33.33
  Week 20 | 0.0 | 66.67 | 58.33
  Week 24 | 0.0 | 58.33 | 58.33
  Week 28 | 0.0 | 58.33 | 58.33
  Week 32 | 0.0 | 41.67 | 41.67

9. Secondary Outcome: Percentage of Participants With 3-point Reduction in QMG Total Score
Description: The percentage of responders with at least a 3-point reduction in QMG total score from baseline is reported. QMG is a physician-reported scale to assess MG disease severity by quantifying several body functions by physical exam. Each question is graded on a 4-point scale from 0=normal to 3=severe with a total score of 0 to 39; the higher score indicates greater disease burden. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: At Weeks 4, 6, 8, 10, 12, 14, 16, 20, 24, 28 and 32
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants
  Week 4 | 25.00 | 50.00 | 16.67
  Week 6 | 16.67 | 41.67 | 33.33
  Week 8 | 33.33 | 66.67 | 33.33
  Week 10 | 33.33 | 66.67 | 33.33
  Week 12 | 41.67 | 75.00 | 25.00
  Week 14 | 33.33 | 66.67 | 25.00
  Week 16 | 33.33 | 58.33 | 33.33
  Week 20 | 0.0 | 41.67 | 33.33
  Week 24 | 0.0 | 41.67 | 33.33
  Week 28 | 0.0 | 41.67 | 25.00
  Week 32 | 0.0 | 16.67 | 16.67

10. Secondary Outcome: Percentage of Participants With 3-point Reduction in MGC Total Score
Description: The percentage of responders with at least a 3-point reduction in MGC total score from baseline is reported. MGC is an assessment scale of MG disease activity based on a combination of participant- and physician-reported items. Items are scored based on 4 potential levels of impact: normal, mild, moderate, or severe with a total score of 0 to 50; the higher score indicates worse MG disease activity. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: At Weeks 4, 6, 8, 10, 12, 14, 16, 20, 24, 28 and 32
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants
  Week 4 | 66.67 | 75.00 | 41.67
  Week 6 | 83.33 | 66.67 | 58.33
  Week 8 | 83.33 | 83.33 | 58.33
  Week 10 | 83.33 | 75.00 | 50.00
  Week 12 | 75.00 | 91.67 | 58.33
  Week 14 | 66.67 | 83.33 | 50.00
  Week 16 | 66.67 | 75.00 | 41.67
  Week 20 | 0.0 | 75.00 | 58.33
  Week 24 | 0.0 | 66.67 | 50.00
  Week 28 | 0.0 | 58.33 | 50.00
  Week 32 | 0.0 | 41.67 | 25.00

ADVERSE EVENTS:
Time Frame: From signing the informed consent form up to end of long-term follow-up (up to Week 32)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | TAK-079 Placebo-matching | TAK-079 300 mg | TAK-079 600 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 8/12 | 9/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-079 Placebo-matching (N=12) | TAK-079 300 mg (N=12) | TAK-079 600 mg (N=12)
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-079 Placebo-matching (N=12) | TAK-079 300 mg (N=12) | TAK-079 600 mg (N=12)
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 1 | 0
Bartholin's abscess (Infections and infestations) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood immunoglobulin A decreased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 3
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Early satiety (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2
Feeling cold (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site haematoma (General disorders) | 1 | 0 | 0
Injection site hypertrophy (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Joint noise (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT04159805/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04159805/SAP_001.pdf